CLINICAL TRIAL: NCT04501705
Title: Clinical Study of Apatinib in the Treatment of Recurrent Atypical/malignant Meningioma in Adults
Brief Title: Apatinib in the Treatment of Recurrent Atypical/malignant Meningioma in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Junping Zhang, professor, Beijing Sanbo Brain Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BJ-CM-Ⅱ-008
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Atypical/malignant Meningioma
MeSH Terms: conditions — Meningioma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- test group (Experimental)
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Apatinib Mesylate — Apatinib mesylate tablets: Orally, 500 mg, once a day, with warm water for half an hour after a meal (the time of taking the medicine every day should be the same as possible).
  Continue to use 28 days as a cycle, medication until disease progression (PD), intolerable toxicity occurs or the patient withdraws informed consent. However, the longest period does not exceed 24 cycles, and the treatment after 24 cycles is determined by the investigator.

SUMMARY:
Apatinib mesylate may be an effective treatment for recurrent atypical/malignant meningioma. This prospective clinical study is now planned to verify the effectiveness and safety of apatinib mesylate in the treatment of relapsed atypical/malignant meningioma.

DETAILED DESCRIPTION:
Vascular endothelial growth factor VEGF is related to the abnormal angiogenesis of meningioma and can also activate other growth factor pathways. Meningiomas are vascular tumors. Studies have shown that the expression of VEGF in atypical meningiomas is twice that of benign meningiomas, and VEGF in anaplastic meningiomas is 10 times that of benign meningiomas. Therefore, anti-angiogenesis therapy may be more effective for higher grade meningiomas. Previous clinical studies have confirmed that anti-angiogenic drugs such as bevacizumab, sunitinib and PTK 787 can slow down tumor growth and prolong progression-free survival for recurrent atypical/malignant meningioma. In summary, apatinib mesylate may be an effective treatment for recurrent atypical/malignant meningioma. This prospective clinical study is now planned to verify the effectiveness and safety of apatinib mesylate in the treatment of relapsed atypical/malignant meningioma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old (at the time of enrollment), regardless of gender.
2. The pathological diagnosis of atypical/malignant meningioma was clear after biopsy or surgery.
3. The tumor recurrence is confirmed by MRI, that is, the diameter of the lesion on the enhanced MRI image is ≥1cm, and ≥2 slices (slice interval 5mm) are visible; or after another biopsy or surgery, the pathological diagnosis is atypical/malignant meningioma.
4. Previous surgery and radiotherapy (including conventional radiotherapy or stereotactic radiosurgery treatment) are required. There are no restrictions on whether to receive chemotherapy or the number of times of the above treatments
5. The time interval from the last radiotherapy is ≥4 weeks.
6. The time interval from the last chemotherapy is ≥4 weeks, and the patients have fully recovered from the acute toxicity of the last treatment.
7. The interval between the last biopsy or surgery is ≥2 weeks.
8. KPS score ≥50 points.
9. If the patient is on glucocorticoid therapy, the hormone dosage has stabilized or decreased for at least 2 weeks before the baseline MRI.
10. The expected survival time is ≥12 weeks.
11. The main organ functions are normal, and there is no serious blood, heart, lung, liver, kidney dysfunction and immune deficiency diseases. The laboratory inspection meets the following requirements:

(1) Routine blood examination, which must be met (no blood transfusion within 14 days):

1. HGB≥100g/L;
2. WBC≥3.0×109/L; NEUT≥1.5×109/L;
3. PLT ≥100×109/L; (2) The biochemical inspection shall meet the following standards:

a. BIL≤1.5 times the upper limit of normal (ULN); b. ALT and AST≤2.0×ULN; c. Serum Cr≤1.5×ULN or endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula); (3) Occult blood in stool (-); (4) Urine routine is normal, or urine protein <(++), or 24-hour urine protein <1.0 g; (5) Left ventricular ejection fraction (LVEF) ≥50%. 12. The coagulation function is normal, without active bleeding and thrombosis.

1. International standardized ratio INR≤1.5×ULN;
2. Partial thromboplastin time APTT≤1.5×ULN;
3. Prothrombin time PT≤1.5ULN. 13. Female patients of childbearing age must undergo a negative pregnancy test (serum or urine) within 7 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of apatinib mesylate tablets ; Male patients of childbearing age should agree to use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of apatinib mesylate tablets.

   14. Patients need to provide 25-30 pieces of tumor tissue slices after the last biopsy or surgery.

   15. The patient has normal swallowing function and can swallow the tablet intact.

   16. The patient voluntarily joined the study and signed an informed consent form (ICF).

   17. The patient is expected to have good compliance and be able to follow up the efficacy and adverse reactions as required by the protocol.

   Exclusion Criteria:
   1. Past application of anti-tumor angiogenesis drugs;
   2. Patients diagnosed with neurofibromatosis type 2 and other tumor syndromes;
   3. People who are known to be allergic to any component of apatinib mesylate;
   4. Antiepileptic drugs that induce liver enzymes are being used, unless antiepileptic drugs that have been replaced with non-hepatic enzymes are at least 2 weeks away from enrollment;
   5. Patients with other malignant tumors, unless they have survived for 5 years and the investigator believes that the risk of recurrence is low or patients with carcinoma in situ;
   6. Patients with hypertension who cannot be reduced to the normal range after treatment with antihypertensive drugs (systolic blood pressure ≤ 140 mmHg / diastolic blood pressure ≤ 90 mmHg);
   7. Patients with coronary heart disease ≥2 grade, arrhythmia (including QTc prolongation in men>450 ms, women>470 ms) and cardiac insufficiency;
   8. Urine routine test indicates urine protein ≥(++), or 24-hour urine protein ≥1.0g;
   9. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5×ULN), have bleeding tendency or are receiving thrombolytic or anticoagulant therapy;
   10. There are many factors that affect the absorption of oral drugs, such as uncontrollable nausea and vomiting, chronic diarrhea and intestinal obstruction;
   11. There is an infection that is difficult to control;
   12. Those who had significant blood coughing up 2 months before enrollment, or had blood volume of 2.5ml or more per day; had clinically significant bleeding symptoms or had clear bleeding tendency within 3 months before enrollment, such as Gastrointestinal bleeding, hemorrhagic gastric ulcer, gastrointestinal perforation, stool occult blood++ and above at baseline, intratumoral or intracranial hemorrhage, or vasculitis, etc.;
   13. Arterial/venous thrombosis events that occurred within 6 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
   14. Pregnant or breast-feeding women; fertility patients who are unwilling or unable to take effective contraceptive measures;
   15. Other situations that the researcher thinks are not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
PFS-6 % | 6-month progression-free survival
  6-month progression-free survival

SECONDARY OUTCOMES:
ORR | up to 5 years
  Objective Response Rate
OS | up to 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Sanbo Brain Hospital, Beijing, Beijing Municipality, China